CLINICAL TRIAL: NCT04192097
Title: Impact of a Curriculum About Professionalism on Stress Response During a Critical Situation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Grenoble Alps (Other)
Responsible Party: Principal Investigator, Pierre ALBALADEJO, Clinical Professor, University Grenoble Alps
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CESAR003
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Professional Burnout; Professional Stress; Anesthesia; Medical Education; High Fidelity Simulation; Anxiety State
Keywords: Cardiopulmonary arrest; Family patient meeting
MeSH Terms: conditions — Burnout, Professional; Occupational Stress; Anxiety Disorders; Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional teaching (No Intervention): No specific curriculum about professionalism
- Professionalism curriculum (Experimental): Traditional teaching + professionalism curriculum
  Interventions: Other: Professionalism curriculum

INTERVENTIONS:
Other: Professionalism curriculum — One year training program including ten two-hours sessions about
  * Knowing yourself
  * Interaction with patients and their families
  * Teamwork and organization with colleagues
  Arms: Professionalism curriculum

SUMMARY:
The purpose of this study is to evaluate the impact of a curriculum about professionalism on stress response during a critical situation in anesthesiology residents. Residents in anesthesiology will complete a training program on professionalism during their first postgraduate year. They will go through a standardized simulated scenario where they have to manage an intra-hospital cardiorespiratory arrest and then meet the patient's family. Stress response will be assessed and compared to a control group that did not receive the training program.

ELIGIBILITY:
Inclusion Criteria:

* Residents in anesthesiology (Postgraduate year 1)
* Voluntary

Exclusion Criteria:

* /

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Psychological stress response : State Trait Anxiety Inventory (STAI) | 1 year
  STAI -State (State-Trait Anxiety Inventory), from 20 to 80, psychological stress response is higher when score is higher

SECONDARY OUTCOMES:
Clinical performance on cardiopulmonary arrest | 1 year
  All simulations will be videotaped and the clinical performance of each participant will be assessed by an independent evaluator using a specific pre-established checklist
Physiological stress response : Standard Deviation | 1 year
  Heart rate variability evaluated by Standard Deviation Normal to Normal, in milliseconds. Physiological stress response is higher when Standard Deviation Normal to Normal, is lower.
Family meeting quality : Gather-Resources-Identify-Educate-Verify-Inquire-"Nuts and bolts"-Give | 1 year
  All simulations will be videotaped and the family meeting quality will be assessed by an independent. Score GRIEV-ING from 0 to 27 evaluator, using the Gather, Resources, Identify, Educate, Verify, Inquire, Nuts and bolts, Give), from 0 to 27, family meeting is better when score is higher
Non technical skills (NTS) : Crisis resource management ( CRM). Score Ottawa | 1 year
  Score Ottawa from 5 to 35
Burnout Scale | 1 year
  Maslach Burnout Inventory, from 0 to 132 points, exploring three dimensions of professional burnout
Quality Of Life : WHOQoL | 1 year
  WHOQoL-8 (World Health Organization Quality of Life), from 12 to 60 points, quality of life is higher when the score is lower
Psychological stress response | 1 year
  Stress Visual Analogical Scale, from 0 to 100, psychological stress response is higher when score is higher

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Grenoble Alps, La Tronche, France

IPD SHARING:
Plan to Share IPD: Undecided